CLINICAL TRIAL: NCT04358653
Title: The Effectiveness of Group Intervention Exercise on Fall Risk Factors Reduction in Community-Dwelling Older Adults
Brief Title: Exercise Effectiveness on Fall Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Garyfallia Pepera, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 118/02-10-2018
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Functionality, Falls, Elderly, Fall Prevention, Exercise Elderly, Assessment, Rehabilitation, Community-Dwelling
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fall prevention exercise program (Experimental): The experimental group was designed to undergo supervised exercise 2 days a week for 8 consecutive weeks for 45-50 min/session. The intervention program was implemented at the nursing home facilities.
  Interventions: Other: fall prevention exercise program
- Control Group (No Intervention): The control group did not receive any intervention during that period and were instructed to pursue their habitual daily life activities.

INTERVENTIONS:
Other: fall prevention exercise program — The intervention protocol was starting with a 10 minute warm up (5 minutes circular walking combined with neck rotation in clockwise and counterclockwise fashion and 5 minutes upper and lower limp stretching exercises) and was followed by 30 minutes of exercises that were aiming to muscle strengthening, balance improvement and functionability enhancement. The muscle strengthening routine consisted of exercises both from standing and sitting position using an elastic band, heel and toe standing, upper limb strengthening using dumbbells. Balance training consisted of standing on one leg, shifting weight laterally from one foot to the other, staggered stance, side stepping. Functionalibility improvement was promoted through walking upstairs and downstairs, standing up from sitting to upright position. At the end a 5 minute cool down procedure was following consisting of circular walking, mild head movements and upper and lower body stretching.
  Other Names: Exercise Rehabilitation; Group exercise program; Physical exercise therapy
  Arms: fall prevention exercise program

SUMMARY:
Objective: To assess the effectiveness of an intervention exercise program on enhancing fall risk deterrent factors, such as balance, postural control, overall strength, functionability in community-dwelling individuals.

Design: Single-blinded randomized controlled trial, comparing two groups, with follow-ups at the begging and 15 days after the completion of the program

Setting: Nursing homes in Ano Volos and Kanalia

Participants: A total of 40 elderly people, both male and female, aged 65 years and older were randomly assigned to an intervention exercise group (n = 20) and a control group (n = 20).

Interventions: Intervention exercise program consisted of two sessions each week for 8 consecutive weeks. The control group received no exercise intervention.

Measurements: Main outcomes were measured by the Timed Up and Go Test, Berg Balance Scale, 10-second chair stand test, Saehan hand grip dynamometer, Upper and Lower Limp reach tests.

DETAILED DESCRIPTION:
Methods Research design

A single - blind, randomized controlled trial design was used to examine the effects of a fall prevention exercise program in reducing fall incidence and fall risks for community-dwelling older adults at a risk for falls. The study was approved by the ethics committee of University of Thessaly.

Sample Forty (40) community dwelling elderly individuals, both males and females, were recruited from nursing homes. Convenience sampling was used. Subject eligibility criteria were: a) 65 years of age and older, b) absence of serious health problems or neurological diseases, c) absence of dementia, d) no recent surgeries. Out of the 40 subjects meeting the above criteria, 20 were randomly assigned to the control group (mean age 79.3±5.49) and 20 to the rehabilitation group (mean age 79.6±7.38). In both groups, 10 subjects reported at least one incidence of falling during the past year whilst the remaining 10 the absence of any.

Base line assessment A structured questionnaire was used to record a) anthropometric and demographic data (age, weight, height, profession etc.), b) comorbid medical conditions (e.g., hypertension, diabetes mellitus, cardiovascular disease, psychiatric illness), c) prescribed medications including psychotropic medications (antidepressants, and sedative hypnotics), d) use of walking aids, e) prior history of falls and fall-related injuries during the past year, f) prior surgeries

Procedure

The experimental group was designed to undergo supervised exercise 2 days a week for 8 consecutive weeks for 45-50 min/session. The intervention program was implemented at the nursing home facilities. The control group did not receive any intervention during that period and were instructed to pursue their habitual daily life activities.

Instruments and assessments (outcome measures) Participants were assessed prior to the beginning of their program and 15 days after the completion of the intervention. Parameters being assessed were: weight, height, BMI, systolic pressure, diastolic pressure, heart rate, grip strength, upper and lower limb force, plus upper and lower extremity elasticity, equilibrium and functionality.

Mobility was assessed using the Time Up & Go Test (TUG) which was measured by recording the time taken to stand up from a standard chair (43cm), walk 3m at a natural pace, turn around, and sit back down in the chair. Expected time for the completion of this task is estimated at 7-10''. (Viccaro et al 2011)

Functional balance was assessed with the Berg Balance Scale that has been developed to measure an elderly person's static and dynamic balancing abilities. It is composed of a total of 14 items and a full score of 56 points. The time required is around 15 minutes. Higher scores indicate better degrees of balance. Based on the total score participants are classified in: a) need for a wheelchair (0-20 points), b) need of aiding tools to walk (21-40 points), c) independent (41 points or higher). Persons with scores of 40 points or higher are not likely to fall (Berg et al., 1992 ; Bogle & Newton 1996; Downs et al 2013)

Grip strength was measured using the SAEHAN hand grip dynamometer. The subject was sitting on a standard chair with the elbow flexed at 900. When the subject was ready, he would begin to strain the device in a maximal isometric effort, maintaining, at the same time, high concentration, as this was a required condition for maximal results. No other body movement was allowed during testing.

Lower Limb's strength was assessed through the "sit to stand 10" trial. Subjects were asked to sit on a chair, stand up and return to the sitting position for 10 consecutive times at full speed, with no intervals between. Normal time expected for the successful completion of the trial was estimated at 24"-27"

Lower Body Flexibility was assessed using a modified Sit and Reach test. This test was performed in a standard chair with one leg fully extended and the other in a flexed position. Participants reached forward with one hand as far as possible and held this position for three seconds. Distance between fingers and toes was measured.

For Upper Body Flexibility assessment, subjects were instructed to bring their hand back as high as possible in order to reach the A7 vertebra. The distance between the thumb and the A7 vertebra was measured (Collins et al 2004) Intervention The intervention protocol was starting with a 10 minute warm up (5 minutes circular walking combined with neck rotation in clockwise and counterclockwise fashion and 5 minutes upper and lower limp stretching exercises) and was followed by 30 minutes of exercises that were aiming to muscle strengthening, balance improvement and functionability enhancement. The muscle strengthening routine consisted of exercises both from standing and sitting position using an elastic band (hip flexion, extension, abduction, adduction, knee flexion and extension, ankle dorsi and plantar flexion), heel and toe standing, upper limb strengthening using dumbbells. Balance training consisted of standing on one leg, shifting weight laterally from one foot to the other, staggered stance, side stepping. Functionalibility improvement was promoted through walking upstairs and downstairs, standing up from sitting to upright position. At the end a 5 minute cool down procedure was following consisting of circular walking, mild head movements and upper and lower body stretching.

Throughout the whole duration of the intervention the elderly subjects were provided with constant feedback for the maintenance of the proper sitting and standing posture.

Breathing rate, blood pressure and heart rate were monitored at every interventional session. All participants were asked to immediately declare any symptom or feeling of dizziness or general discomfort and on that case the current intervention would stop.

ELIGIBILITY:
Inclusion Criteria:

Community-Dwelling Older Adults >65 years old

Exclusion Criteria:

* absence of neurological diseases
* absence of dementia
* no recent surgeries.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Mobility | 8 weeks
  Mobility was assessed using the Time Up & Go Test (TUG) which was measured by recording the time taken to stand up from a standard chair (43cm), walk 3m at a natural pace, turn around, and sit back down in the chair. Expected time for the completion of this task is estimated at 7-10''. (Viccaro et al 2011)
Functional balance | 8 weeks
  Functional balance was assessed with the Berg Balance Scale that has been developed to measure an elderly person's static and dynamic balancing abilities. It is composed of a total of 14 items and a full score of 56 points. The time required is around 15 minutes. Higher scores indicate better degrees of balance. Based on the total score participants are classified in: a) need for a wheelchair (0-20 points), b) need of aiding tools to walk (21-40 points), c) independent (41 points or higher). Persons with scores of 40 points or higher are not likely to fall (Berg et al., 1992 ; Bogle & Newton 1996; Downs et al 2013)
Upper Limb Strength | 8 weeks
  Upper Limb Strength was measured using the SAEHAN hand grip dynamometer. The subject was sitting on a standard chair with the elbow flexed at 900. When the subject was ready, he would begin to strain the device in a maximal isometric effort, maintaining, at the same time, high concentration, as this was a required condition for maximal results. No other body movement was allowed during testing.
Lower Limb strength | 8 weeks
  Lower Limb's strength was assessed through the "sit to stand 10" trial. Subjects were asked to sit on a chair, stand up and return to the sitting position for 10 consecutive times at full speed, with no intervals between. Normal time expected for the successful completion of the trial was estimated at 24"-27"
Upper Body Flexibility | 8 weeks
  Upper Body Flexibility assessment, subjects were instructed to bring their hand back as high as possible in order to reach the A7 vertebra. The distance between the thumb and the A7 vertebra was measured (Collins et al 2004)
Lower Body Flexibility | 8 weeks
  Lower Body Flexibility was assessed using a modified Sit and Reach test. This test was performed in a standard chair with one leg fully extended and the other in a flexed position. Participants reached forward with one hand as far as possible and held this position for three seconds. Distance between fingers and toes was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Greece

IPD SHARING:
Plan to Share IPD: No